CLINICAL TRIAL: NCT02783196
Title: Advantages of Liraglutide Mediated Through Its Effect on Clock Gene mRNA Expression
Brief Title: Effect of Liraglutide on Clock Genes
Acronym: LIR-CG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0100-16 WOMC
Record Dates: First submitted 2016-05-20; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (LIR) (Experimental): Type 2 diabetic randomized to start with two 40 days treatment periods starting with Liraglutide ( IR) treatment, and then after 2 weeks of wash-out, will crossover to second treatment period of 40 days with placebo (PLA)
  Interventions: Drug: Liraglutide
- Placebo (PLA) (Placebo Comparator): Type 2 diabetic randomized to start with two 40 days treatment periods starting with placebo ( PLA) treatment, and then after 2 weeks of wash-out, will crossover to second treatment period of 40 days with Liraglutide ( LIR)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — In the LIR arm, the participants will be provided with instructions in using pre-filled single-use plastic syringes ready for once daily subcutaneous injection of LIR. From day 1 to day 10, with LIR daily dose of 0.6 mg (0.1 ml), followed by other 10 day courses (from day 11 to day 20) with LIR 1.2 mg (0.2 ml), then will be up-titrated to high dose 1.8 mg (0.3 ml) of LIR (from day 21 to day 40). At crossover-day 40, the participants will undergo a 14 days wash-out period, day 41 to day 55.
  Other Names: LIR
  Arms: Liraglutide (LIR)
Drug: Placebo — In the PLA arm, the participants will be provided with instructions in using pre-filled single-use plastic syringes ready for once daily subcutaneous injection of PLA. Will start with PLA with matched volume saline injections of 0.1 ml PLA during the first 10 days, followed by 10 days, with 0.2 ml PLA, thereafter PLA will be up-titrated to highest volume 0.3 ml placebo for the rest of the PLA treatment period . At crossover-day 40, the participants will undergo a 14 days wash-out period, day 41 to day 55.
  Other Names: PLA
  Arms: Placebo (PLA)

SUMMARY:
This study is undertaken to search whether glucagon-like peptide-1 (GLP-1) analogue, Liraglutide, by enhancing clock gene and AMPK-SIRT-1 mRNA expression, may reverse the metabolic abnormalities of type 2 diabetes, improving overall glycemic excursion, inflammatory cytokines and β-cell function in type 2 diabetes individuals.

The investigators aim is to compare the effect of 40 days treatment with Liraglutide (LIR) vs. 40 days with placebo (PLA) in T2D participants on the following end points:

Primary end-points:

* Change in the oscillation of CG (i.e. CLOCK, BMAL1, Per1, Per2, Cry1, Cry2, Rev-erb-alpha Ror-alpha), AMPK, SIRT1 and inflammatory cytokines mRNA expression in white blood cells (WBCs).

Secondary end-points:

* Overall daily glycemic variation assessed with continuous glucose monitoring system (CBMS)
* Serum levels of inflammatory cytokines (TNF-α, IL-1β, IL-6)
* β-Cell function derived from glucose and insulin response to OGTT

DETAILED DESCRIPTION:
Background: Cumulative evidence strongly implicates that the disruption of clock genes (CGs) plays a causative role in insulin resistance, hyperglycemia and β-cell dysfunction in type 2 diabetes (T2D). CGs are synchronized by meal timing. Indeed, in animals and patients with T2D, restricting feeding to specific hours, such as large meals assigned to breakfast with reduced dinner, can reset and restore CG expression, resulting in improved glycemic control, insulin sensitivity and reduction of HbA1c compared to isocaloric diet with a different meal timing (small breakfast and overeating at dinner). Since glucagon-like peptide-1 (GLP-1) is secreted within a few minutes in response to food ingestion and it influences multiple humoral and neural signaling pathways that may further influence CG expression in many cells, it has been suggested that GLP-1 may be a resetting signal for the CGs, synchronizing the food entrainment on CGs expression thereby influencing the glucose metabolism. In fact, several studies in animal models, documented that GLP-1 analogs either exenatide or liraglutide, via activation of CG expression and AMPK-SIRT-1 pathway, improved insulin sensitivity, muscular glucose uptake, reduced hepatic and cardiac steatosis, inflammatory cytokines and oxidative stress, and enhanced β-cell insulin secretion and proliferation, independently of the GLP-1 analog glucose-lowering effects.

To the best of the investigators knowledge, no systemic study in humans to date has investigated the changes in the expression of CGs and AMPK-SIRT-1 pathway, concomitantly with the effect on glycemic control, insulin sensitivity, beta cell function, and inflammatory cytokines in T2D individuals during treatment with Liraglutide or other GLP-1 analogs.

Hypothesis: The investigators hypothesize, that Liraglutide, by enhancing CG and AMPK-SIRT-1 expression may reverse the metabolic abnormalities of T2D, improving insulin sensitivity, overall glycemic excursion, inflammatory cytokines and β-cell function in T2D individuals.

Objectives:

The investigators aim is to compare the effect of 40 days treatment with Liraglutide (LIR) vs. 40 days with placebo (PLA) in T2D participants on the following end points:

Primary end-points:

* Change in the oscillation of CG (i.e. CLOCK, BMAL1, Per1, Per2, Cry1, Cry2, Rev-erb-alpha, Ror-alpha), AMPK, SIRT1 and inflammatory cytokines mRNA expression in white blood cells (WBCs).

Secondary end-points:

* Overall daily glycemic variation assessed with continuous glucose monitoring system (CBMS)
* Serum levels of inflammatory cytokines (TNF-α, IL-1β, IL-6)
* β-Cell function derived from glucose and insulin response to OGTT

Methods: In a randomized, double blind crossover-within-subject clinical trial, the investigators will study 18 weight- matched obese and overweight participants with known T2D, diagnosed < 20 years, and HbA1c 7.0 to 10 %, BMI: 26-32 kg/m2 treated with diet alone or diet plus metformin, and sodium/glucose cotransporter 2 (SGLT2) inhibitors (gliflozins).

All 18 T2D participant will undergo randomization at baseline to two 40 days treatment periods, either starting with LIR treatment, and then after 2 weeks of wash-out, will crossover to second treatment period of 40 days with PLA, or vice-versa, starting the first period with PLA during 40 days and then crossover to 40 days with LIR. The treatment with LIR and PLA will be up-titrated progressively from 0.1ml to 0.3ml to avoid the secondary effects of LIR.

Expected results: The investigators expect that LIR will lead to enhanced expression of the diurnal oscillation of the CGs and AMPK, SIRT1 pathway, will reduce serum inflammatory cytokines, and overall daily glycemic variation while improving insulin sensitivity and β-Cell function.

Significance of the study: Showing that GLP-1 analog Liraglutide, improves β-cell function in type 2 diabetic individuals, by enhancing clock genes mRNA expression and the AMPK-SRIT1 pathway, may change the approach of Liraglutide treatment, from being an excellent anti-diabetic agent with beneficial effect on the diabetic heart, to a drug with the ability to synchronize body metabolism and improve glucose homeostasis in health and disease. Presently, there are many available drugs for the treatment of type 2 diabetes, but their mode of action does not make any of them more advantageous. If this GLP-1 analog not only reduces glucose, body weight and cardiovascular risk, but also synchronizes the circadian clock, this would make of Liraglutide the drug of choice (immediately after metformin) for the treatment of obesity, early diabetes and for prevention of T2D complications and cardiovascular events in high risk patients, moreover, Liraglutide by influencing clock genes expression, may further prevent several other age related disorders linked to the disruption of clock genes.

ELIGIBILITY:
Inclusion Criteria

1. Patients with T2D diagnosed that were diagnosed < 20 years.
2. HbA1c: 7 to 10 % at screening and at qualification
3. BMI: 26-32 kg/m2.
4. Men and women
5. Between the ages of 30 and 75 years.
6. Patients treated with diet alone or diet plus metformin and SGLT2 inhibitors, at a stable dose for at least 3 months.
7. Concomitant medication i.e. antihypertensive, anti-lipidemic, anti-thrombotic drugs will be allowed.
8. Patients that usually wake up between 06:00 and 07:00 and go to sleep between 22:00 and 24:00.
9. Subjects should not have shift work within 6 month of the study and should not have crossed time zones within 1 month of the study.
10. For woman of child bearing potential, negative pregnancy test and willingness to use birth control during the study :

Exclusion Criteria:

1. Type 1 diabetes or secondary forms of diabetes.
2. Use of glucose-lowering therapy apart from metformin and SGLT2 inhibitors.
3. Treatment with GLP-1 receptor agonists, dipeptidyl peptidase-4 (DPP-4) inhibitors within the last 3 months.
4. Major illness with life expectancy < 5 years.
5. Serum creatinine level >2mg/d or renal dysfunction: (estimated glomerular filtration rate <45 mL/min/1.73 m2).
6. Hepatic dysfunction: liver disease or transaminase levels >3-fold above normal.
7. History of acute or chronic pancreatitis or high risk for pancreatitis i.e. triglycerides over 400 mg/dl or alcoholism.
8. Family or personal history of Multiple Endocrine Neoplasia type 2 (MEN-2) or familial medullary thyroid carcinoma.
9. Familial or personal history of multiple endocrine neoplasia type 2 (MEN2), familial or non-familial medullary thyroid carcinoma (MTC)
10. Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer).
11. Those taking psychotropic, anorectic medication, steroid treatment or with illicit drug abuse or alcoholism within one year prior to study onset.
12. Congestive heart failure and all cardiac arrhythmias i.e. atrial fibrillation.
13. Pregnancy or lactation.
14. Eating disorders and subjects after bariatric surgery or affected by gastroparesis.
15. Night or rotating shift workers or those who crossed more than 2 time zones during the 2-week period prior to study onset.
16. No change in medication or nutrition supplements or physical activity will be made during the study period.
17. Known proliferative retinopathy or maculopathy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clock Gene expression | Up to 95 days
  The Clock Genes mRNA expression will be assessed in white blood cells

SECONDARY OUTCOMES:
AMPK mRNA expression | Up to 95 days
  he AMPK mRNA expression will be assessed in white blood cells on day 0, on day 40 and on day 95
SIRT1 mRNA expression | Up to 95 days
  SIRT1 mRNA expression will be assessed in white blood cells on day 0, on day 40 and on day 95
Beta-cell function | Up to 92 days
  Beta-cell function based on oral glucose tolerance test (OGTT) will be assessed on day -3, on day 37 and on day 92
Overall glycemia | Up to 95 days
  Overall glycemia assessed with continuous glucose monitoring system (CGMS) will be performed during 3 days at baseline from day - 3 to day 0, again from day 37 to 40 and three days before the end of intervention from day 92 to day 95

CONTACTS AND LOCATIONS:
Overall Officials: Julio Wainstein, MD, Principal Investigator — Diabetes Unit Wolfson Medical center
Locations (1):
- Diabetes Unit E. Wolfson Hospital, Holon, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No